CLINICAL TRIAL: NCT01291862
Title: Obstructive Sleep Apnea, Retinal Vein Occlusion, Retinal Artery Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-2010-0008
Record Dates: First submitted 2011-02-01; First posted 2011-02-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Retinal Vascular Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Watchpat 100 — Watchpat 100 is a noninvasive portable sleep monitoring device which monitors peripheral arterial tone, pulse, oxygen saturation, snoring, and body position. Patient places one probe at his or her finger and another sensor at front of the chest and Watchpat 100 monitors the patient overnight.
  Other Names: Watch-PAT™ 100

SUMMARY:
Obstructive sleep apnea is a common disorder linked to serious long-term adverse health consequences; such as hypertension, metabolic dysfunction, cardiovascular disease. Retinal vascular occlusion is related to many systemic illnesses especially hypertension. Obstructive sleep apnea is also related to vascular endothelial dysfunction and vascular endothelial growth factor elevation which causes vision threatening complications of retinal vascular occlusion. Therefore the relationship between obstructive sleep apnea and retinal vascular occlusion should be studied.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who visits outpatient clinic and diagnosed as retinal vascular occlusion which occurred within recent 3 months

Exclusion Criteria:

* Any ocular disease other than retinal vascular occlusion (for example: floppy eyelid syndrome, uveitis, glaucoma, other retinal diseases)
* Patient who has difficulty answering the questionnaires or portable sleep monitoring
* Patient who refuses the study enroll

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Watchpat-100(noninvasive portable sleep monitoring device) | after finishing the tests with Watchpat-100
  Result Data of Watchpat-100 : apnea-hypopnea index(AHI)
Berlin questionnaire | after finishing the Berlin questionnaire
  Incidence of patients at risk for obstructive sleep apnea according to the Berlin questionnaire
Epworth sleepiness scale | after finishing the Epworth sleepiness sclae
  Incidence of patients with daytime sleepiness according to the Epworth sleepiness scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kwon HJ, Kang EC, Lee J, Han J, Song WK. Obstructive Sleep Apnea in Patients with Branch Retinal Vein Occlusion: A Preliminary Study. Korean J Ophthalmol. 2016 Apr;30(2):121-6. doi: 10.3341/kjo.2016.30.2.121. Epub 2016 Mar 25. PMID 27051260